CLINICAL TRIAL: NCT01519518
Title: A Randomised Controlled Trial to Compare Unfractionated Heparin Versus Bivalirudin in the Treatment of Patients With a Clinical Diagnosis of ST-Segment Elevation Myocardial Infarction Events - For Planned Management With Primary PCI
Brief Title: How Effective Are Antithrombotic Therapies in Primary Percutaneous Coronary Intervention
Acronym: HEAT-PPCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Rod Stables, Consultant Cardiologist, Liverpool Heart and Chest Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 923
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-04

CONDITIONS: Acute ST Elevation Myocardial Infarction
Keywords: ST elevation myocardial infarction; Primary percutaneous coronary intervention; Unfractionated heparin; Bivalirudin; primary angioplasty
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Heparin; bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unfractionated heparin (Active Comparator): 70 units/kg body weight intravenous
  Interventions: Drug: unfractionated heparin
- bivalirudin (Active Comparator): intravenous bolus of 0.75 mg/kg followed by infusion of 1.75 mg/kg per hour
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: unfractionated heparin — 70 units/kg body weight intravenous
  Other Names: UFH
  Arms: Unfractionated heparin
Drug: Bivalirudin — intravenous bolus of 0.75 mg/kg followed by infusion of 1.75 mg/kg per hour
  Other Names: Angiox
  Arms: bivalirudin

SUMMARY:
The purpose of this study is to compare unfractionated heparin (UFH) and bivalirudin in the performance and subsequent outcomes of Primary percutaneous coronary intervention. This will be a pragmatic trial. Interventional procedures will be performed to reflect current and evolving standards, including predominant radial access. All patients will be treated with routine oral anti-platelet therapy pre-procedure. GP IIb/IIIa inhibitors will be reserved for 'bail out' treatment only.

DETAILED DESCRIPTION:
HEAT-PPCI is a single-centre prospective, dual-arm, open-label, randomised controlled trial comparing two antithrombotic agents in patients undergoing PPCI. All patients presenting to the PPCI service at Liverpool Heart and Chest Hospital will be assessed for trial eligibility. The patients will be allocated by randomisation in equal proportions to the two treatment groups receiving UFH (70 units/kg prior to the procedure) or bivalirudin (bolus of 0.75 mg/kg prior to the start of the intervention, followed by an infusion of 1.75 mg/kg per hour for the duration of the procedure).

Pre-Specified Subgroup Analyses

* Subgroup analyses looking at the impact of access site comparing radial versus femoral route
* Assessment of the outcomes in diabetic patients receiving oral hypoglycaemic or insulin therapy versus all other patients
* Comparing the outcomes in patients < or ≥ 75 years of age
* Type of p2y12 receptor inhibiting antiplatelet agent (Examples: clopidogrel, prasugrel, ticagrelor)
* Patients with impaired LV function versus normal LV function
* Patients managed with actual or attempted primary PCI versus no immediate PCI procedure attempted

PLATELET FUNCTION SUBSTUDY A substudy will be performed to assess indices of coagulation and platelet function studies comparing the impact of heparin or bivalirudin therapy on coagulation status at the end of the PPCI procedure. This study will be performed on all patients treated between the hours of 0800 and 1600, Monday to Friday. A single blood sample taken at the time of general blood sampling for routine clinical screening will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting with a suspected myocardial infarction event with PPCI as the proposed index reperfusion strategy will be included in the trial

Exclusion Criteria:

* ≤ 18 years of age
* Known intolerance, hypersensitivity or contraindication to any trial medication
* Active bleeding at presentation
* Artificial ventilation, reduced conscious level or other factors precluding the administration of oral antiplatelet therapy
* Previous enrolment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1829 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rod Stables, MA DM FRCP, Principal Investigator — Liverpool Heart and Chest Hospital, Liverpool, UK
Locations (1):
- Liverpool Heart and Chest Hospital, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Derived] Shahzad A, Kemp I, Mars C, Wilson K, Roome C, Cooper R, Andron M, Appleby C, Fisher M, Khand A, Kunadian B, Mills JD, Morris JL, Morrison WL, Munir S, Palmer ND, Perry RA, Ramsdale DR, Velavan P, Stables RH; HEAT-PPCI trial investigators. Unfractionated heparin versus bivalirudin in primary percutaneous coronary intervention (HEAT-PPCI): an open-label, single centre, randomised controlled trial. Lancet. 2014 Nov 22;384(9957):1849-1858. doi: 10.1016/S0140-6736(14)60924-7. Epub 2014 Jul 4. PMID 25002178
- [Derived] Malik N, Gershlick AH. The clinical and economic impact of bivalirudin for percutaneous coronary intervention. Expert Rev Pharmacoecon Outcomes Res. 2013 Dec;13(6):699-706. doi: 10.1586/14737167.2013.844650. PMID 24219045

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unfractionated Heparin | Bivalirudin
Started | 914 | 915
Completed | 907 | 905
Not Completed | 7 | 10
Not completed — Consent not available | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unfractionated Heparin | Bivalirudin | Total
Number analyzed (Participants) | 907 | 905 | 1812
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.6 [54.0 to 73.8] | 62.9 [53.7 to 74] | 63.2 [53.9 to 73.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 258 | 502
  Male | 663 | 647 | 1310

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac Events (MACE) in Terms of the Incidence of All Cause Mortality, Cerebrovascular Accident, Re-infarction and Additional Unplanned Target Lesion Revascularization
Time Frame: 28 days
Measure: Number; unit: percentage of total participants
Arm/Group | Unfractionated Heparin | Bivalirudin
Number analyzed (Participants) | 907 | 905
percentage of total participants | 5.7 | 8.7

2. Primary Outcome: Type 3-5 Bleeding According to BARC (Bleeding Academic Research Consortium)Definition
Time Frame: 28 days
Measure: Number; unit: percentage of total participants
Arm/Group | Unfractionated Heparin | Bivalirudin
Number analyzed (Participants) | 907 | 905
percentage of total participants | 3.1 | 3.5

3. Secondary Outcome: CKMB Release Following Index Revascularisation Measured With a Single Estimation 12-18 Hours After the Procedure
Time Frame: 28 days
Reporting Status: Not Posted

4. Secondary Outcome: Minor Bleeding: Type 2 Bleeding According to BARC (Bleeding Academic Research Consortium) Definition
Time Frame: 28 days
Measure: Number; unit: percentage of total participants
Arm/Group | Unfractionated Heparin | Bivalirudin
Number analyzed (Participants) | 907 | 905
percentage of total participants | 10.8 | 9.2

5. Secondary Outcome: Stent Thrombosis Rate (ARC Definite or Probable)
Time Frame: 28 days
Measure: Number; unit: percentage of total participants
Arm/Group | Unfractionated Heparin | Bivalirudin
Number analyzed (Participants) | 907 | 905
percentage of total participants | 0.9 | 3.4

6. Secondary Outcome: For Illustration, and to Allow Comparison With Existing Trials the Rate of Net Adverse Clinical Events (NACE), Combining the Primary Safety and Efficacy Outcomes
Time Frame: 28 days
Reporting Status: Not Posted

7. Secondary Outcome: All Cause Mortality
Time Frame: 1 year
Reporting Status: Not Posted

8. Secondary Outcome: Development of Thrombocytopenia
Time Frame: 28 days
Reporting Status: Not Posted

9. Secondary Outcome: Door-to-first Device Time
Time Frame: 28 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Unfractionated Heparin | Bivalirudin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No